CLINICAL TRIAL: NCT03241017
Title: A Phase II Trial Investigating the Benefit of Immunotherapy With Durvalumab After Autologous Transplant in High-risk Diffuse-large B-cell Lymphomas (the IDA-D Trial)
Brief Title: Durvalumab in DLBCL After Autologous Transplant
Acronym: IDA-D
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Celgene withdrew the support for this study (Durvalumab cannot be provided)
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDA-D Trial
Record Dates: First submitted 2017-07-26; First posted 2017-08-07 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: Diffuse Large B-Cell Lymphoma; Double-hit Lymphomas; Grey Zone Lymphomas; Double or Triple Expressor Lymphomas; Unclassifiable Aggressive Lymphoma types; Aggressive Lymphomas
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, single-center, open-label, single-arm, non-comparative and non-randomized phase II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab (Experimental): Durvalumab 1500 mg (day 1) given every 4 weeks for a total of 12 applications (1 year).
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Immunotherapy with Durvalumab after ASCT

SUMMARY:
The trial assess the progression-free survival (PFS) two years after autologous stem cell transplantation (ASCT) in high-risk DLBCL patients receiving PD-L1 inhibition with durvalumab.

DETAILED DESCRIPTION:
Background and Rationale:

Autologous stem cell transplantation (ASCT) is standard of care in the treatment concept of adult patients with multiple myeloma (MM), malignant lymphomas (including diffuse large B-cell lymphomas (DLBCL), mantle cell lymphomas, follicular lymphomas or T-cell lymphomas), acute myeloid leukemia (AML) and relapsing germ cell tumors. The number of patients treated with ASCT is steadily increasing, e.g. by +17% alone in Switzerland in the year 2015, to a total of 464 ASCT per year in Switzerland. The Inselspital (University Hospital) in Berne is the leading hospital in Switzerland for ASCT, with 145 ASCT in the year 2015. Among these 145 transplants, 31 patients had DLBCL.

The goal of treatment in DLBCL is definite cure. In DLBCL, the addition of anti-CD20 treatment to standard CHOP (Cyclophosphamid, Doxorubicin, Vincristine, Prednisone) chemotherapy has improved the cure rate after R-CHOP (Rituximab-CHOP) first-line treatment. Nevertheless, the disease is relapsing in roughly 20% of these patients. At relapse, patients are treated with salvage chemotherapy such as the R-DHAP (Rituximab, Dexamethasone, Cisplatin,Cytarabine), or R-ICE (Rituximab,Ifosfamide, Carboplatin, Etoposide) regimens, followed by BEAM (BCNU, Etoposide, Cytarabine, Melphalan) or BeEAM (Bendamustin, Etoposide, Cyclophosphamide, Melphalan) high-dose chemotherapy supported with ASCT. The overall survival rate at the Inselspital Bern and elsewhere at two years for DLBCL patients after ASCT is 60%, and, therefore, improving outcome of such patients remains an unmet clinical need. This is particularly true in high-risk DLBCL patients, such as in DLBCL patients relapsing within 12 months after first-line treatment as well as in DLBCL patients not achieving a (first or second) complete remission (CR) after induction treatment before ASCT. PFS at two years for such high-risk lymphoma patients is 50% at the investigators' institution.

Immunotherapy (such as with PD-L1 inhibition) after ASCT is a promising approach to potentially improve results after ASCT. A first study applying PD-1 inhibition with three applications (every 42 days) of Pidilizumab started between days 30 and 90 after ASCT showed a promising progression-free survival rate of 72% in relapsing DLBCL patients at 16 months after the first Pidilizumab application. These data suggest that immunotherapy after ASCT has the potential to a meaningful improvement of survival rates in DLBCL patients after ASCT.

Objective:

The primary objective of this Trial is to show a progression-free survival of 70% two years after autologous stem cell transplantation (ASCT) in high-risk DLBCL patients receiving PD-L1 inhibition with durvalumab.

Study Duration:

The 46 patients needed in this study will be included within 24 months. Additional 24 months will be needed until the last study patient reaches PFS at 2 years. Accordingly, the total study duration is expected to be 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any types of DLBCL (de novo or transformed), including double-hit lymphomas, grey zone lymphomas, double or triple expressor lymphomas, unclassifiable aggressive lymphoma types or aggressive lymphomas.
* Lymphoma patients (as listed above) in first remission considered as high-risk and defined as lymphoma patients not achieving a complete first remission after induction treatment before subsequent ASCT; or patients in second remission considered as high-risk and defined as lymphoma patients relapsing within 12 months after first-line treatment or lymphoma patients not achieving a complete second remission after salvage treatment before subsequent ASCT.
* ECOG 0-2
* Age 18-75 years
* Female patients of child-bearing potential must have a negative pregnancy test (urine or serum) within 14 days prior to study treatment, and they must implement adequate measures (hormonal treatment p.o. or i.m., intra uterine surgical devices, or latex condoms) to avoid pregnancy during study treatment and for additional 12 months.
* Patients must have given voluntary written informed consent.

Exclusion Criteria:

* Other types of malignant lymphomas
* Previous treatment with antibodies against PD-(L)1
* Symptomatic CNS (Central Nervous System) involvement by lymphoma
* Active infection requiring antibiotic/antifungal treatment
* Lack of patient cooperation to allow study treatment as outlined in this protocol
* Pregnancy or lactating female patients
* Major surgery less than 30 days before start of treatment
* Contraindications and hypersensitivity to any of the active chemotherapy compounds

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 24 months
  Number of Patients with Progression-free survival (PFS) two years after autologous stem cell transplantation (ASCT) in high-risk DLBCL patients receiving PD-L1 inhibition with durvalumab.

SECONDARY OUTCOMES:
Response Rate | 24 months
  The Response (Tumor measurement) to durvalumab treatment will be assessed by PET-CT 24 months after ASCT
Adverse Events | 24 months
  Number of Patients experiencing Toxicity (Adverse Events)
Hematologic engraftment | 24 months
  Number of days until hematological engraftment. Hematologic engraftment after high-dose chemotherapy induced myelosuppression is defined as the first day of neutrophils rising again above 0.5 G/l, and of platelets rising again above 20 G/L in the absence of platelet transfusions in the previous 3 days. Hematological values will be performed every 4 weeks
The quality of life | 24 months
  The EORTC Q30 questionnaire will be given to patients before the first durvalumab administration, and after 3, 12 and 24 months after ASCT to assess quality of life.
Overall Survival | 24 months
  Number of Patient alive at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pabst, MD, Study Chair — Departement of Medical Oncology, University Hospital Berne